CLINICAL TRIAL: NCT01912924
Title: A Prospective Single Centre Open Label Trial to Assess the Effectiveness of the Use of Spinal Cord Stimulation in Subjects With Chronic Knee Pain "Failed Knee Surgery"
Brief Title: A Prospective Trial for the Effectiveness of the Use of Spinal Cord Stimulation (SCS) in Failed Knee Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult enrollment, no subjects identified to enroll
Sponsor: Coastal Orthopedics & Sports Medicine (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGFK001
Record Dates: First submitted 2010-02-03; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Pain
Keywords: chronic pain from failed knee surgery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spinal cord stimulator (Boston Scientific) — spinal cord stimulator trial leads and hand held battery
  Other Names: Boston Scientific

SUMMARY:
A study for patients who have chronic postoperative pain who had knee replacement surgery. If qualified, a 14 day trial and an implantation of spinal cord stimulator for control of pain will be administered. This study will evaluate effectiveness of pain control. Subjects will be followed for one year post implantation.

DETAILED DESCRIPTION:
Male and Female over the age of 18 who have had a total knee replacement at least nine months ago. Continue with unilateral knee pain equal to or greater than 4 on a 1 to 10 scale. Subjects will receive a trial placement of spinal cord stimulator for 5 to 10 days. if trial is successful subjects will proceed to permanent placement of stimulator for the treatment of the knee pain. subjects will then be followed post implant to assess the effectiveness of the stimulator for the pain.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* total knee replacement at least nine months prior to enrollment
* unilateral knee pain at least 4 or more on a 1-10 visual analog scale
* failed other conservative treatments -

Exclusion Criteria:

* life expectancy of at least 6 months
* significant disease including Complex Regional Pain Syndrome,ipsilateral radiculopathy
* presence of pacemaker/vns or other Spinal Cord Stimulator
* previous lumbar surgery
* active infection
* unable to hold anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | one year
  standardized visual pain scale

SECONDARY OUTCOMES:
Health Related Quality of Life | one year
  Health Related Quality of Life standardized questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Gennady Gekht, MD, Principal Investigator — Coastal Orthopedics & Sports Medicine
Locations (1):
- Coastal Orthopedics & Sports Medicine, Bradenton, Florida, United States